CLINICAL TRIAL: NCT07109349
Title: Effect of Transcutaneous Auricular Neurostimulation on Mental Wellness and Resiliency for First Responders: A Pilot Trial
Brief Title: tAN for First Responders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spark Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBM-MRES-01
Record Dates: First submitted 2025-07-30; First posted 2025-08-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Mental Fatigue; Mental Stress
Keywords: Mental resilience; tAN; Transcutaneous Auricular Neurostimulation; Vagus nerve stimulation; Neurostimulation; First responders; taVNS; Police officer
MeSH Terms: conditions — Mental Fatigue; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Active tAN (Experimental): First responders will self-administer once-daily active tAN sessions for 1-2 hours for 28 days. Participants will complete daily and weekly assessments to evaluate levels of stress, mood, energy/fatigue, sleep quality , and burnout. Daily assessments and tAN sessions will cease after Day 28. Participants will continue to complete weekly assessments until Day 56.
  Interventions: Device: Sparrow Link

INTERVENTIONS:
Device: Sparrow Link — Sparrow Link will be using the components of the Sparrow Ascent device: (FDA-cleared K230796) a wearable, battery-operated, neurostimulation system designed to transcutaneously stimulate nerves on and/or around the auricle. Participants will self-administer daily active tAN sessions on Days 1 - 28.
  Other Names: Transcutaneous Auricular Neurostimulation

SUMMARY:
This study is designed as an open label, single arm, decentralized clinical study in which first responders will receive transcutaneous auricular neurostimulation (tAN), which targets the auricular branch of the vagus nerve (ABVN) via the mastoid and the auriculotemporal nerve (ATN) anterior to the tragus. Participants will be enrolled in the study over the course of eight weeks (56 days).

Participants will respond to daily and weekly questionnaires regarding mood, stress, sleep, energy/fatigue, and burnout. Each week, participants will complete consolidated online questionnaires (intended to last no longer than 15 minutes) comprised of the Perceived Stress Short-Form (PSS-4), Well-Being Index (WHO-5), Mini-Z Burnout (5-item), PROMS Sleep Disturbance (PROMIS-SD), GAD-7 (every 2 weeks), and Perceived Stress (PSS-10; monthly). The PSS-10 will replace the PSS-4 on Days 0, 28, and 56.

No tAN treatment will be delivered during the Baseline Period (days between Study Introduction and Day 0). Participants will complete the weekly set of questionnaires ("Weekly Questionnaires") on Day 0. Participants will be recommended to complete the daily set of questionnaires ("Daily Questionnaires ") on the other days of the Baseline Period.

On Days 1 - 28, participants will self-administer one session of one to two hours of tAN therapy each day. Participants will be recommended to complete the daily tAN session post-shift prior to sleep. Weekly Questionnaires will be completed by participants on Study Days 0, 7, 14, 21, 28, 35, 42, 49, and 56. Participants will be recommended to complete Daily Questionnaires on all other study days, up to Day 28. Daily Questionnaires will not be required to be completed by participants. Daily tAN sessions and Daily Questionnaires will cease after Day 28. Participants will complete a Study Satisfaction Questionnaire with the Weekly Questionnaires on Day 56.

Following Day 56, participants will schedule a Study Exit Interview with the Research Coordinator.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is currently employed in a first responder position
2. Age ≥ 18 years
3. Reliable access to an internet-enabled device to complete required questionnaires
4. GAD-7 score ≥ 5

Exclusion Criteria:

1. Participant has a history of epileptic seizures
2. Participant has a history of neurologic diseases or traumatic brain injury
3. Participant has presence of devices (e.g., pacemakers, cochlear prostheses or implants, neurostimulators)
4. Participant has abnormal left ear anatomy or ear infection present
5. Participant has auditory impairment of the left ear (ruptured eardrum, deafness, tinnitus, etc.)
6. Participant is currently enrolled in another interventional trial
7. Women of childbearing potential, not using adequate contraception as per the investigator's judgement
8. Females who are pregnant or lactating
9. Participant has any other significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-07-10 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
GAD-7 | Screening, Day 0, Day 14, Day 28, Day 42, Day 56
  The GAD-7 is a valid and efficient tool for screening for GAD and assessing its severity in clinical practice and research. The questionnaire consists of 7 questions in which participants are asked to rate each item on a 0 (not at all) to 3 (nearly every day). GAD-7 total score for the seven items ranges from 0 to 21 where 0-4 represents minimal anxiety, 5-9 represents mild anxiety, 10-14 represents moderate anxiety and 15-21 represent severe anxiety.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS-4, PSS-10) | Weekly throughout enrollment beginning Day 0 through Day 56)
  The PSS-4 is a brief version of the Perceived Stress Scale used to assess the degree to which situations in one's life are appraised as stressful. The questionnaire consists of 4 items, with participants rating each on a 0 (never) to 4 (very often) scale. Scores range from 0 to 16, with higher scores indicating greater perceived stress. The PSS-10 consists of 10 items that assess how unpredictable, uncontrollable, and overloaded respondents find their lives. Each item is rated on a 0 (never) to 4 (very often) scale. Total scores range from 0 to 40, with higher scores indicating greater perceived stress.
  The PSS-10 will replace the PSS-4 on Days 0, 28, and 56.
PROMIS Sleep Disturbance | Weekly throughout enrollment beginning Day 0 through Day 56)
  The PROMIS Sleep Disturbance measure evaluates self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. Participants respond to 8 items rated on a 1 (not at all) to 5 (very much) scale. Raw scores are converted to T-scores with a mean of 50 and a standard deviation of 10, where higher scores indicate greater sleep disturbance. The tool is suitable for use in clinical and research populations.
WHO-5 Well-Being Index | Weekly throughout enrollment beginning Day 0 through Day 56)
  The WHO-5 is a short, validated measure of current mental well-being. The questionnaire consists of 5 positively worded items rated on a 0 (at no time) to 5 (all of the time) scale. The raw score ranges from 0 to 25 and is multiplied by 4 to yield a final score from 0 to 100, with higher scores indicating greater well-being. A score below 50 suggests reduced well-being and may indicate the need for further assessment.
Mini-Z Burnout Survey | Weekly throughout enrollment beginning Day 0 through Day 56)
  The Mini-Z Burnout Survey is a brief tool for assessing burnout and job satisfaction. It includes 10 items covering emotional exhaustion, stress, satisfaction, and workload. Most items are rated on a 1 to 5 Likert scale. Higher scores on the burnout item (typically scored 1 to 5) reflect greater burnout, with a score of 3 or higher suggesting at least some level of burnout.

CONTACTS AND LOCATIONS:
Overall Officials: Navid Khodaparast, PhD, Principal Investigator — Spark Biomedical, Inc.
Locations (1):
- Spark Biomedical - DECENTRALIZED STUDY, Dallas, Texas, United States